CLINICAL TRIAL: NCT03918616
Title: P2X7 Receptor, Inflammation and Pathophysiology of Neurodegenerative Diseases
Brief Title: P2X7 Receptor, Inflammation and Neurodegenerative Diseases
Acronym: NeuroInfiam
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Anna Solini, Associate Professor, University of Pisa
Other Study IDs: AS0002
Record Dates: First submitted 2019-04-10; First posted 2019-04-17 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Neuro-Degenerative Disease
Keywords: Alzheimer disease; Parkinson disease; P2X7 receptor
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease | interventions — Memantine; Dopamine Agonists; sirio

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD + AD: Patients with newly-diagnosed (onset of suggestive symptoms not later than 3 months) Parkinson disease (PD) or Alzheimer disease (AD) with no previous specific treatment, no anti-inflammatory drugs assumed in the three months preceding the enrolment and no chronic inflammatory diseases or cancer.
  Interventions: Drug: Memantine, Dopamine receptor-agonists
- Control group: An age and gender matched control group (n=50) was formed, on a volunteer basis, by the spouse of the probands participating in the study.

INTERVENTIONS:
Drug: Memantine, Dopamine receptor-agonists — The study do not provide any experimental drugs. Patientes will receive treatment routinary used by Neurologist for these diseases.
  Other Names: Memantine: Ebixa. Dopamine receptor-agonists: Sinemet, Sirio.
  Groups: PD + AD

SUMMARY:
Parkinson disease (PD) is a chronic degenerative disease characterized by a progressive loss of dopaminergic neurons in the substantia nigra. Its pathophysiological mechanisms are still partially unknown; a main role seems to be played by chronic neuroinflammation. A few reports have addressed the possible involvement of the inflammasome in PD, just describing the protective effect of P2X7 purinergic receptor (P2X7R) blockers in murine models of the disease and in microglial cells, where NLRP3 is activated by α-Synuclein, triggering a neuroinflammation that contributes to degeneration of dopaminergic neurons. It is still unclear whether, in addition to the increased brain expression and function of the nucleotide-binding domain, leucine-rich repeat, pyrin domain containing type 3 (NLRP3) inflammasome platform, a systemic activation of such complex might participate in the pathogenesis of PD, which could be the role of the P2X7R in this scenario, and whether such patterns undergo any specific epigenetic regulation. The present study has been designed to address these issues.

DETAILED DESCRIPTION:
The day of the study patientes underwent a complete clinical evaluation and assessment of psycho-physical abilities using specific test such as Mini-Mental State Examination (MMSE), Cognitive Alzheimer's Disease Assessment Scale (ADAS-Cog), Clinical Dementia Rating Scale, Unified Parkinson's Disease Rating Scale (UPDRS). Blood samples were collected from an antecubital vein to assess serum and plasma aliquots for blood routine analysis and RNA and protein extraction from circulating lymphomonocytes.

To explore a putative epigenetic regulation of such complex scenario some circulating miRNAs likely involved in the pathogenesis of neurological diseases and neuro-inflammation will be measured.

Expression and functional activity of P2X7R-inflammasome complex will be measured by PCR and WB. Acute phase cytokines inflammasome-related levels will be determined by ELISA. Biochemical parameters (fasting glucose, lipid profile, serum creatinine, uric acid) will be measured by standard methods in the biochemistry laboratory of the University Hospital in Pisa. The same determinations will be repeated after one year from the first visit.

ELIGIBILITY:
Inclusion Criteria:

* newly-diagnosed PD or AD;
* no previous specific treatment;
* no systemic inflammatory or immunological disease and/or cancer;
* no anti-inflammatory drugs assumed in the three months preceding the enrolment;
* patients able to consent.

Exclusion Criteria:

* history of strokes or any neurological disease;
* patients assuming neuroleptic drugs;
* atypical symptoms at onset.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study consecutively enrolled 50 newly-diagnosed, treatment-naive PD or AD individuals among those referring to the Neurology Unit, University Hospital in Pisa, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in P2X7R-inflammasome activity | each patient will be assessed one year after diagnosis
  NLRP3-ASC-Caspase-1 activity is measured using RT-PCR
Change from baseline in NFkB activity | each patient will be assessed one year after diagnosis
  NFkB activity is measured using RT-PCR
Change from baseline in serum α-synuclein | each patient will be assessed one year after diagnosis
  Circulating levels of α-synuclein are determined using high sensitivity Quantikine enzyme-linked immunosorbent assay (ELISA) and express as [ng/ml]
Change from baseline in serum IL-1β | each patient will be assessed one year after diagnosis
  Circulating levels of IL-1β are determined using high sensitivity Quantikine enzyme-linked immunosorbent assay (ELISA) and express as [pg/ml]
Change from baseline in serum IL-18 | each patient will be assessed one year after diagnosis
  Circulating levels of IL-18 are determined using high sensitivity Quantikine enzyme-linked immunosorbent assay (ELISA) and express as [pg/ml]
Change from baseline in circulating levels of microRNA miR-30 and miR-7 | each patient will be assessed one year after diagnosis
  Circulating levels of microRNA miR-30 and miR-7 are measured using TaqMan Advanced MicroRNA Assays

CONTACTS AND LOCATIONS:
Overall Officials: Anna Solini, MD, PhD, Principal Investigator — Univeristy of Pisa
Locations (1):
- University of Pisa, Pisa, Italy